CLINICAL TRIAL: NCT04183777
Title: Assessment of the Age, Reasons, Oral Health Status and Dental Treatment Needs of Children in Their First Dental Visit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, aya abd el mawgoud mohamed elsanhouri, princile investigator, Cairo University
Other Study IDs: Cairo university ,Egypt
Record Dates: First submitted 2019-11-26; First posted 2019-12-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-12

CONDITIONS: Dental Caries; Parents; Parenting; Pain
Keywords: first dental visit; oral health; reasons of first dental visit; dental treatment needs
MeSH Terms: conditions — Dental Caries; Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to asses the age, reasons, oral health status and dental treatment needs of children in their first dental visit.

DETAILED DESCRIPTION:
We are going to provide each parent or guardian whose children fulfilling the inclusion criteria attending to Department of Paediatrics Dentistry at Cairo University to fulfil questionnaire which include multiple MCQ questions. The state of oral health and dental treatment needs will be assessed based on clinical examination, according to recommendations of the World Health Organization. The total number of teeth and number of teeth affected by decay (d, D) in every child will be recorded. The intensity of caries will be estimated based on the average dmf/DMF number, i.e. caries intensity index.

The dental treatment needs of each child will be assessed based on the following categories:

1. None: no restorative treatment required.
2. Simple: preventive treatment required, such as scaling and brushing, oral hygiene instruction (OHI), application of topical fluoride and fissure sealant.
3. Moderate: one or more of teeth require one or two surface restoration.
4. Complex: one or more teeth require three or four surface restoration / stainless steel crown, endodontic therapy and crown, and /or extraction(7) .

Reasons for first dental visit will be categories as :

a. Adaptive visit dental check-up preventive purpose. b. Tooth pain. c. Emergency case (tooth injury, abscess, infection). d. Decay noted by parent.

e. Any Other. We will explain to the parents and legal guardians the aim of the study without any guiding to prevent any information bias which may occur. The questionnaire will be given before the treatment and will be collected after it. Any children whose records will include missing information will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Children with Primary and mixed dentition.
* Children visiting the dentist for the first time (first dental visit

Exclusion Criteria:

* Children with systemic diseases or physical and mental problem.
* Children whose parents refuse participation

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We are going to provide each parent or guardian whose children fulfilling the inclusion criteria attending to Department of Paediatrics Dentistry at Cairo University to fulfil questionnaire which include multiple MCQ questions. We will explain to the parents and legal guardians the aim of the study without any guiding to prevent any information bias which may occur. The questionnaire will be given before the treatment and will be collected after it. Any children whose records will include missing information will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
reasons for the first dental visit. | 1 year
  There are different reasons for the first dental visit these reasons may be due to a- Adaptive visit dental check-up preventive purpose. b. Tooth pain. c. Emergency case (tooth injury, abscess, infection). d. Decay noted by parent.
  e. Any Other.
  Caregiver will be asked to fill a questionnaire include multiple reasons. The parents or Guardian select the most chief complain for coming to the first dental visit. And after selection the most common reason will determine.

SECONDARY OUTCOMES:
age | 1 years
  Caregiver will be asked to fill a questionnaire include multiple age. The parents or Guardian select the most optimal age for the first dental visit from their point of view .
oral health | 1 years
  The state of oral health will be assessed based on clinical examination, according to recommendations of the World Health Organization. The total number of teeth and number of teeth affected by decay (d, D) in every child will be recorded. The intensity of caries will be estimated based on the average dmf/DMF number, i.e. caries intensity index.
dental treatment needs | 1 years
  Dental treatment needs will be assessed based on clinical examination, according to recommendations of the World Health Organization.
  The dental treatment needs of each child will be assessed based on the following categories:
  1. None: no restorative treatment required.
  2. Simple: preventive treatment required, such as scaling and brushing, oral hygiene instruction (OHI), application of topical fluoride and fissure sealant.
  3. Moderate: one or more of teeth require one or two surface restoration. D-Complex: one or more teeth require three or four surface restoration / stainless steel crown, endodontic therapy and crown, and /or extraction.

CONTACTS AND LOCATIONS:
Overall Officials: aya elsnhouri, bachelor, Principal Investigator — Cairo University
Locations (1):
- Aya Abdelmawgoud Elsanhouri, El-Sheikh Zayed City, Giza Governorate, Egypt